CLINICAL TRIAL: NCT00754741
Title: Phase III Clinical Trial of the Effectiveness of Adherence Data and Motivational Interviewing to Improve Medication Adherence and Both Glycated Hemoglobin and Cholesterol Control
Brief Title: Multi-arm Intervention Diabetes Adherence Study
Acronym: MIDAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, keoki williams, Senior Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DK64695; R01DK064695 (NIH); 5R01DK064695-06 (NIH)
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes
Keywords: medication adherence; motivational interviewing
MeSH Terms: conditions — Diabetes Mellitus; Medication Adherence | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual care (No Intervention): All Physicians are given limited training in how to intervene on poor adherence, but no patient adherence information is provided to these clinicians via electronic prescribing software when they see patients assigned to this arm
- Adherence (Active Comparator)
  Interventions: Behavioral: Adherence information
- Adherence Plus (Active Comparator)
  Interventions: Behavioral: Adherence information plus motivational interviewing

INTERVENTIONS:
Behavioral: Adherence information — Physicians, of the patients randomized to this arm, will have medication adherence information displayed when using the electronic prescribing system.
  Arms: Adherence
Behavioral: Adherence information plus motivational interviewing — Physicians, of the patients randomized to this arm, will have medication adherence information displayed when using the electronic prescribing system. Moreover, patients randomized to this arm will be recruited into a clinic run by pharmacists and nurses with delegated prescription power. The clinic personnel will use motivational interviewing techniques with patients to improve adherence to medications and/or to intensify medical treatment if adherence is optimal.
  Arms: Adherence Plus

SUMMARY:
The purpose of this study is to compare the effectiveness of two different interventions to improve adherence to diabetes medications among patients with diabetes and poor metabolic control.

DETAILED DESCRIPTION:
Nonadherence to medications is common among patients with diabetes and contributes to suboptimal control of glycemic and lipid plasma levels. Adherence is not routinely measured in clinical practice because no valid, feasible methods have been readily available. The lack of medication adherence information contributes to clinician failure to identify and address patient nonadherence and to clinical inertia and poor health outcomes.

Existing electronic prescribing systems hold the potential to display medication adherence information. We propose a 3-arm randomized clinical trial to test the effectiveness of providing primary care physicians (PCPs) with both adherence measurements and an adherence clinic to improve adherence to diabetic and lipid-lowering drugs. This adherence clinic will consist of a pharmacist and nurse trained in motivational interviewing (Ml) techniques to improve adherence to medications.

Adherence indices will be generated by linking e-prescribing information with pharmacy data. The trial will be conducted among 1,436 patients with diabetes and poor blood glycemic and/or lipid control. Patients will be randomized to one of the following three study arms: 1) Usual care - PCPs will write prescriptions electronically but will not be provided patient adherence information or Ml support; 2) Intervention - PCPs will be provided adherence information and prompts electronically when using the electronic prescribing system; and 3) Intervention - PCPs will be provided adherence information and prompts electronically when using the electronic prescribing system plus physicians and patients will receive support from an adherence clinic.

Our intervention uses as theoretical behavioral framework elements of the Chronic Care Model, Self-Determination Theory, and the Health Belief Model. The study will use qualitative methods to guide intervention design and implementation and will include both process evaluation and treatment fidelity measures. The intervention will be tailored to patients' adherence and goal levels. The study will also evaluate the cost effectiveness of the intervention. Patients will be followed for 36 months. The introduction of sustainable medication adherence monitoring in clinical practice holds great potential to improve health outcomes among patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 dispensings for oral medications used to treat diabetes and dyslipidemia in the last 18 month.
* At least one laboratory result for both glycated hemoglobin and LDL-cholesterol in the last 6 months.
* Average HbA1c ≥ 7% OR an average LDL ≥ 100 mg/d
* Continuous health plan enrollment currently and in the previous calendar year with no more than a 1 month lapse of coverage, and benefits that include both medical and pharmacy coverage.

Exclusion Criteria:

* Patients who have been institutionalized in a nursing home or in a long-term care facility for more than 3 months in the preceding 18 month period.
* Participation in a disease management program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1692 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janis Campbell, RN, Study Director — Henry Ford Health System; Manel Pladeval, MD, MS, Principal Investigator — Henry Ford Hospital; L. Keoki Williams, MD, MPH, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Background] Pladevall M, Williams LK, Potts LA, Divine G, Xi H, Lafata JE. Clinical outcomes and adherence to medications measured by claims data in patients with diabetes. Diabetes Care. 2004 Dec;27(12):2800-5. doi: 10.2337/diacare.27.12.2800. PMID 15562188
- [Background] Heisler M, Hogan MM, Hofer TP, Schmittdiel JA, Pladevall M, Kerr EA. When more is not better: treatment intensification among hypertensive patients with poor medication adherence. Circulation. 2008 Jun 3;117(22):2884-92. doi: 10.1161/CIRCULATIONAHA.107.724104. Epub 2008 May 27. PMID 18506011
- [Background] Schmittdiel JA, Uratsu CS, Karter AJ, Heisler M, Subramanian U, Mangione CM, Selby JV. Why don't diabetes patients achieve recommended risk factor targets? Poor adherence versus lack of treatment intensification. J Gen Intern Med. 2008 May;23(5):588-94. doi: 10.1007/s11606-008-0554-8. Epub 2008 Mar 4. PMID 18317847
- [Background] Choudhry NK, Patrick AR, Antman EM, Avorn J, Shrank WH. Cost-effectiveness of providing full drug coverage to increase medication adherence in post-myocardial infarction Medicare beneficiaries. Circulation. 2008 Mar 11;117(10):1261-8. doi: 10.1161/CIRCULATIONAHA.107.735605. Epub 2008 Feb 19. PMID 18285564
- [Background] Ho PM, Magid DJ, Shetterly SM, Olson KL, Peterson PN, Masoudi FA, Rumsfeld JS. Importance of therapy intensification and medication nonadherence for blood pressure control in patients with coronary disease. Arch Intern Med. 2008 Feb 11;168(3):271-6. doi: 10.1001/archinternmed.2007.72. PMID 18268167
- [Background] Odegard PS, Capoccia K. Medication taking and diabetes: a systematic review of the literature. Diabetes Educ. 2007 Nov-Dec;33(6):1014-29; discussion 1030-1. doi: 10.1177/0145721707308407. PMID 18057270
- [Background] Williams LK, Joseph CL, Peterson EL, Wells K, Wang M, Chowdhry VK, Walsh M, Campbell J, Rand CS, Apter AJ, Lanfear DE, Tunceli K, Pladevall M. Patients with asthma who do not fill their inhaled corticosteroids: a study of primary nonadherence. J Allergy Clin Immunol. 2007 Nov;120(5):1153-9. doi: 10.1016/j.jaci.2007.08.020. Epub 2007 Oct 22. PMID 17936894
- [Background] Piette JD. Interactive behavior change technology to support diabetes self-management: where do we stand? Diabetes Care. 2007 Oct;30(10):2425-32. doi: 10.2337/dc07-1046. Epub 2007 Jun 22. No abstract available. PMID 17586735
- [Background] Borrelli B, Riekert KA, Weinstein A, Rathier L. Brief motivational interviewing as a clinical strategy to promote asthma medication adherence. J Allergy Clin Immunol. 2007 Nov;120(5):1023-30. doi: 10.1016/j.jaci.2007.08.017. Epub 2007 Sep 29. PMID 17904625
- [Background] West DS, DiLillo V, Bursac Z, Gore SA, Greene PG. Motivational interviewing improves weight loss in women with type 2 diabetes. Diabetes Care. 2007 May;30(5):1081-7. doi: 10.2337/dc06-1966. Epub 2007 Mar 2. PMID 17337504
- [Background] Munro S, Lewin S, Swart T, Volmink J. A review of health behaviour theories: how useful are these for developing interventions to promote long-term medication adherence for TB and HIV/AIDS? BMC Public Health. 2007 Jun 11;7:104. doi: 10.1186/1471-2458-7-104. PMID 17561997
- [Background] Channon SJ, Huws-Thomas MV, Rollnick S, Hood K, Cannings-John RL, Rogers C, Gregory JW. A multicenter randomized controlled trial of motivational interviewing in teenagers with diabetes. Diabetes Care. 2007 Jun;30(6):1390-5. doi: 10.2337/dc06-2260. Epub 2007 Mar 10. PMID 17351283
- [Background] van Dulmen S, Sluijs E, van Dijk L, de Ridder D, Heerdink R, Bensing J. Patient adherence to medical treatment: a review of reviews. BMC Health Serv Res. 2007 Apr 17;7:55. doi: 10.1186/1472-6963-7-55. PMID 17439645
- [Background] Grant R, Adams AS, Trinacty CM, Zhang F, Kleinman K, Soumerai SB, Meigs JB, Ross-Degnan D. Relationship between patient medication adherence and subsequent clinical inertia in type 2 diabetes glycemic management. Diabetes Care. 2007 Apr;30(4):807-12. doi: 10.2337/dc06-2170. Epub 2007 Jan 26. PMID 17259469
- [Background] Williams LK, Joseph CL, Peterson EL, Moon C, Xi H, Krajenta R, Johnson R, Wells K, Booza JC, Tunceli K, Lafata JE, Johnson CC, Ownby DR, Enberg R, Pladevall M. Race-ethnicity, crime, and other factors associated with adherence to inhaled corticosteroids. J Allergy Clin Immunol. 2007 Jan;119(1):168-75. doi: 10.1016/j.jaci.2006.09.029. Epub 2006 Nov 2. PMID 17208598
- [Background] Ho PM, Rumsfeld JS, Masoudi FA, McClure DL, Plomondon ME, Steiner JF, Magid DJ. Effect of medication nonadherence on hospitalization and mortality among patients with diabetes mellitus. Arch Intern Med. 2006 Sep 25;166(17):1836-41. doi: 10.1001/archinte.166.17.1836. PMID 17000939
- [Background] Miller NH, Hill M, Kottke T, Ockene IS. The multilevel compliance challenge: recommendations for a call to action. A statement for healthcare professionals. Circulation. 1997 Feb 18;95(4):1085-90. doi: 10.1161/01.cir.95.4.1085. PMID 9054774
- [Background] Haynes RB, Ackloo E, Sahota N, McDonald HP, Yao X. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD000011. doi: 10.1002/14651858.CD000011.pub3. PMID 18425859

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Started | 567 | 569 | 556
Completed | 510 | 500 | 502
Not Completed | 57 | 69 | 54
Not completed — Died or disenrolled | 57 | 69 | 54

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing | Total
Number analyzed (Participants) | 567 | 569 | 556 | 1692
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (11.5) | 63.3 (10.9) | 64.5 (10.5) | 64.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302 | 270 | 266 | 838
  Male | 265 | 299 | 290 | 854
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 224 | 237 | 238 | 699
  White | 297 | 294 | 281 | 872
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 46 | 38 | 37 | 121
HbA1c [Mean (Standard Deviation); unit: %] | 8.0 (1.4) | 8.2 (1.4) | 8.0 (1.3) | 8.0 (1.4)
LDL-C [Mean (Standard Deviation); unit: mg/dL] | 99.9 (31.4) | 98.5 (33.8) | 97.1 (31.5) | 98.5 (32.2)
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.1 (0.4) | 1.1 (0.3) | 1.2 (0.9) | 1.1 (0.6)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 133.6 (15.4) | 132.3 (15.3) | 133.2 (15.8) | 133.0 (15.5)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 74.8 (10.0) | 75.6 (9.3) | 75.0 (9.2) | 75.1 (9.5)
Insulin use [Number; unit: participants] | 187 | 191 | 192 | 570
Biguanide use [Number; unit: participants] | 335 | 364 | 347 | 1046
Thiazolidinedione use [Number; unit: participants] | 78 | 85 | 73 | 236
Sulfonylurea use [Number; unit: participants] | 327 | 341 | 337 | 1005
Alpha-glucosidase inhibitor use [Number; unit: participants] | 5 | 4 | 3 | 12
Meglitinide use [Number; unit: participants] | 8 | 3 | 2 | 13
Statin use [Number; unit: participants] | 446 | 452 | 443 | 1341
Ezetimibe use [Number; unit: participants] | 73 | 77 | 90 | 240
Fibrate use [Number; unit: participants] | 59 | 51 | 50 | 160
Niacin use [Number; unit: participants] | 7 | 6 | 5 | 18
Bile acid sequestrant use [Number; unit: participants] | 9 | 4 | 3 | 16
Oral diabetes medication adherence [Mean (Standard Deviation); unit: Adherence - proportion] — Adherence is the estimated proportion of the prescribed dose taken over a 3-month period. Therefore, each estimate of medication adherence represented a 3-month window of use prior to and including the assessment time (e.g., the adherence estimate at baseline represented use beginning 3 months before randomization and ending at the time of randomization). Pharmacy claims data (i.e., days supply and refill frequency) were used to estimate adherence.
  Adherence - proportion | 0.76 (0.35) | 0.76 (0.35) | 0.75 (0.36) | 0.75 (0.36)
Lipid-lowering medication adherence [Mean (Standard Deviation); unit: Adherence - proportion] — Adherence is the estimated proportion of the prescribed dose taken over a 3-month period. Therefore, each estimate of medication adherence represented a 3-month window of use prior to and including the assessment time (e.g., the adherence estimate at baseline represented use beginning 3 months before randomization and ending at the time of randomization). Pharmacy claims data (i.e., days supply and refill frequency) were used to estimate adherence.
  Adherence - proportion | 0.71 (0.37) | 0.70 (0.37) | 0.69 (0.37) | 0.70 (0.37)

OUTCOME MEASURES:

1. Primary Outcome: Glycated Hemoglobin Levels
Time Frame: at 18 months post randomization
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 569 | 556
Percent | 7.88 (1.53) | 7.91 (1.53) | 7.79 (1.34)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.763, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.285, ANOVA

2. Primary Outcome: LDL-cholesterol Levels
Time Frame: at 18 months post randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 569 | 556
mg/dL | 89.02 (32.11) | 87.27 (35.67) | 85.56 (32.86)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.380, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.084, ANOVA

3. Secondary Outcome: Adherence to Oral Anti-diabetic Medications
Description: Adherence is the estimated proportion of the prescribed dose taken over a 3-month period. Therefore, each estimate of medication adherence represented a 3-month window of use prior to and including the endpoint time (e.g., the adherence estimate at "6 months post randomization" represented use beginning at 3 months post-randomization and ending at 6 months post-randomization). Pharmacy claims data (i.e., days supply and refill frequency) were used to estimate adherence at each endpoint date.
Time Frame: at 6 months post randomization
Measure: Mean (Standard Deviation); unit: Adherence - proportion
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 569 | 556
Adherence - proportion | 0.75 (0.35) | 0.74 (0.36) | 0.74 (0.37)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.667, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.530, ANOVA

4. Secondary Outcome: Adherence to Lipid-lowering Drugs
Description: as for outcome 3
Time Frame: at 6 months post randomization
Measure: Mean (Standard Deviation); unit: Adherence - proportion
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 569 | 556
Adherence - proportion | 0.70 (0.37) | 0.69 (0.36) | 0.69 (0.36)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.881, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.849, ANOVA

5. Secondary Outcome: Cardiovascular Morbidity and Mortality (Exploratory)
Time Frame: at 24 months post randomization
Measure: Number; unit: participants
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 568 | 556
participants | 63 | 80 | 58
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.134, Chi-squared
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.714, Chi-squared

6. Secondary Outcome: Glycated Hemoglobin Levels
Time Frame: at 6 months post randomization
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 569 | 556
Percent | 7.81 (1.42) | 7.90 (1.44) | 7.81 (1.41)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.291, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.968, ANOVA

7. Secondary Outcome: LDL Cholesterol Levels
Time Frame: at 6 months post randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 568 | 556
mg/dL | 92.92 (32.33) | 92.07 (36.68) | 91.23 (31.17)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.671, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.399, ANOVA

8. Secondary Outcome: Glycated Hemoglobin Levels
Time Frame: at 12 months post randomization
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 569 | 556
Percent | 7.94 (1.60) | 7.96 (1.54) | 7.84 (1.40)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.829, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.283, ANOVA

9. Secondary Outcome: LDL Cholesterol Levels
Time Frame: at 12 months post randomization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 569 | 556
mg/dL | 90.63 (32.41) | 90.70 (36.90) | 87.43 (32.43)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.971, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.115, ANOVA

10. Secondary Outcome: Adherence to Oral Anti-diabetic Medications
Description: Adherence is the estimated proportion of the prescribed dose taken over a 3-month period. Therefore, each estimate of medication adherence represented a 3-month window of use prior to and including the endpoint time (e.g., the adherence estimate at "12 months post randomization" represented use beginning at 9 months post-randomization and ending at 12 months post-randomization). Pharmacy claims data (i.e., days supply and refill frequency) were used to estimate adherence at each endpoint date.
Time Frame: at 12 months post randomization
Measure: Mean (Standard Deviation); unit: Adherence - proportion
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 569 | 556
Adherence - proportion | 0.75 (0.35) | 0.74 (0.36) | 0.74 (0.38)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.573, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.443, ANOVA

11. Secondary Outcome: Adherence to Oral Anti-diabetic Medications
Description: Adherence is the estimated proportion of the prescribed dose taken over a 3-month period. Therefore, each estimate of medication adherence represented a 3-month window of use prior to and including the endpoint time (e.g., the adherence estimate at "18 months post randomization" represented use beginning at 15 months post-randomization and ending at 18 months post-randomization). Pharmacy claims data (i.e., days supply and refill frequency) were used to estimate adherence at each endpoint date.
Time Frame: at 18 months post randomization
Measure: Mean (Standard Deviation); unit: Adherence - proportion
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 567 | 556
Adherence - proportion | 0.75 (0.36) | 0.73 (0.37) | 0.73 (0.38)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.469, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.369, ANOVA

12. Secondary Outcome: Adherence to Lipid-lowering Drugs
Description: as for outcome 10
Time Frame: at 12 months post randomization
Measure: Mean (Standard Deviation); unit: Adherence - proportion
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 569 | 556
Adherence - proportion | 0.70 (0.36) | 0.69 (0.37) | 0.69 (0.37)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.779, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.733, ANOVA

13. Secondary Outcome: Adherence to Lipid-lowering Drugs
Description: as for outcome 11
Time Frame: at 18 months post randomization
Measure: Mean (Standard Deviation); unit: Adherence - proportion
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 569 | 556
Adherence - proportion | 0.70 (0.37) | 0.70 (0.37) | 0.70 (0.37)
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.952, ANOVA
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.856, ANOVA

14. Secondary Outcome: Cardiovascular Morbidity and Mortality (Exploratory)
Time Frame: at 36 months post randomization
Measure: Number; unit: participants
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Number analyzed (Participants) | 567 | 569 | 556
participants | 101 | 112 | 99
Statistical Analysis 1: Comparison: Usual Care vs Adherence Information; Test type: Superiority or Other; p = 0.419, Chi-squared
Statistical Analysis 2: Comparison: Usual Care vs Adherence Information Plus Motivational Interviewing; Test type: Superiority or Other; p = 0.998, Chi-squared

ADVERSE EVENTS:
Arm/Group | Usual Care | Adherence Information | Adherence Information Plus Motivational Interviewing
Serious Adverse Events (participants affected / at risk) | 0/567 | 0/569 | 0/556
Other Adverse Events (participants affected / at risk) | 0/567 | 0/569 | 0/556

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No